CLINICAL TRIAL: NCT04191811
Title: Moment-to-moment Neural Variability as a Predictor of Treatment Outcome in Patients With Common Psychiatric Disorders: Major Depressive Disorder, Insomnia and Social Anxiety Disorder
Brief Title: Investigating Neural Response Variability as a Single-patient Predictor of Successful CBT in Clinical Psychiatry
Acronym: TreVar
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristoffer N T Månsson, Principal Investigator, Karolinska Institutet
Other Study IDs: 2021-06396-0
Record Dates: First submitted 2019-12-02; First posted 2019-12-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-03

CONDITIONS: Psychiatric Disorder; Depression; Anxiety Disorders; Insomnia
Keywords: Internet-delivered Cognitive Behavior Therapy; BOLD-fMRI; Moment-to-moment variability
MeSH Terms: conditions — Mental Disorders; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Depression Internet-delivered CBT: 12 weeks of guided internet-delivered CBT for depression.
  Interventions: Behavioral: Internet-delivered cognitive behavioral therapy for major depressive disorder
- Insomnia Internet-delivered CBT: 12 weeks of guided internet-delivered CBT for insomnia.
  Interventions: Behavioral: Internet-delivered cognitive behavioral therapy for insomnia
- Social Anxiety Internet-delivered CBT: 12 weeks of guided internet-delivered CBT for social anxiety.
  Interventions: Behavioral: Internet-delivered cognitive behavioral therapy for social anxiety disorder

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behavioral therapy for major depressive disorder — Cognitive behavioral therapy delivered over a period of 12 weeks, guided by a psychologist who provides written feedback on home assignments and questions.
  Groups: Depression Internet-delivered CBT
Behavioral: Internet-delivered cognitive behavioral therapy for insomnia — Cognitive behavioral therapy delivered over a period of 12 weeks, guided by a psychologist who provides written feedback on home assignments and questions.
  Groups: Insomnia Internet-delivered CBT
Behavioral: Internet-delivered cognitive behavioral therapy for social anxiety disorder — Cognitive behavioral therapy delivered over a period of 12 weeks, guided by a psychologist who provides written feedback on home assignments and questions.
  Groups: Social Anxiety Internet-delivered CBT

SUMMARY:
Many psychiatric patients are not sufficiently improved by current interventions. Functional magnetic imaging brain imaging (fMRI) has proven to be a promising method for predicting treatment outcomes in psychiatric treatment. Individuals moment-to-moment variability have not yet been evaluated as a predictor of treatment of three common forms of mental illness: depression, insomnia and health anxiety. The goal is to investigate whether objective measurements of brain function contribute to a better prediction of a patient's success in treatment than experiences and self-reports, e.g., treatment credibility and patients expectations about the treatment. The prediction model will be tested on internet-delivered CBT (iCBT) for depression, insomnia and social anxiety. Patients in each diagnostic group are asked for participation before treatment. The total number of participants in this study will amount to 225 participants. The goal is that 35% consists of healthy controls and that the remaining part is equally distributed between the three diagnostic patient groups.

Being able to better predict how well a psychiatric treatment will work for an individual has great value from both an economic and a treatment perspective. The findings from this study may contribute to increased knowledge about neurobiological complications in mental illness. In the longer term, it can lead to improved routines and help in clinical decision-making when patients should be recommended treatment.

DETAILED DESCRIPTION:
Background: There is extensive evidence that cognitive behavioral therapy (CBT) is an effective method of treating common psychiatric disorders such as depression, social anxiety and insomnia. However, access to CBT is very limited. Furthermore, evidence suggest that internet-delivered CBT (iCBT) is as effective as traditional CBT. However, many psychiatric patients are not sufficiently improved by current interventions. Functional brain imaging has proven to be a promising method for predicting treatment outcomes in psychiatric treatment. Calculations on brain signal variability based on the blood-oxygen-level-dependent, BOLD signal (BOLD-fMRI) is a relatively new technique, shown to accurately predict chronological age and cognitive performance. Preliminary data from the investigators' lab suggest that pre-treatment BOLD-fMRI variability is predictive of CBT outcome in patients with social anxiety disorder.

Objectives: The objective of the study is to investigate whether objective measurements of brain function, in comparison with subjective experiences and self-reports (e.g., rating on treatment credibility and patients expectations about the treatment), contribute to better prediction of treatment outcome. The prediction model will be tested on iCBT for three common forms of mental disorders (depression, insomnia and social anxiety). Furthermore, participants will be compared with healthy controls to better understand neurobiological factors that may contribute to mental illness. Preliminary data from the investigators' lab suggest that BOLD-fMRI variability differs between social anxiety disorder participants and healthy individuals.

Method: A sample of outpatients scheduled for iCBT treatment for depression, insomnia or social anxiety at the Internet Psychiatry Unit at Karolinska University Hospital in Huddinge, Stockholm, will be invited to participate in the study. In addition to clinical participants, a healthy control group will be recruited via advertisement in social media. The length of the iCBT intervention is 12 weeks, during which participants engage in web-based treatment modules in a sequential manner, guided though a digital messaging system by a licensed psychologist who provides support and feedback on progress and assignments.

Measuring instruments: Brain imaging is performed before the patients initiate psychiatric treatment. The brain will be examined with structural and functional magnetic resonance imaging (MRI) using an EPI sequence to capture the BOLD signal (Philips 3-Tesla, 32 channel head-coil).

During the online self-referral process and during clinical intake interview, data on a number of potential predictor variables are collected:

* Within the social-demographic domain: age; gender; relationship status (dichotomized as being single or not); level of education rated on a 7-point scale (1 = less than 7-9 years in school; 2 = 7-9 years in school; 3 = incomplete vocational or secondary school; 4 = vocational school; 5 = secondary school; 6 = university, started but not completed studies; 7 = completed university studies); employment status dichotomized as working full-time or not; having children, living situation (alone, with kids, with partner, other), if they do physical activity weekly or not, if they smoke or not.
* Within the clinical characteristics domain: duration of illness (years since onset), history of psychotropic medication, if currently on psychotropic medication, history of inpatient psychiatric care, history of depression and attempted suicide, presence of a neuropsychiatric diagnosis (e.g. ADHD or autism spectrum disorder), current or previous psychological treatment and current or previous periods of sick leave.
* Presence (yes/no) of any comorbid illness is assessed using the the MINI-International Neuropsychiatric Interview (MINI), including bipolar disorder, panic disorder, agoraphobia, social anxiety disorder, mild depressive episode, moderate depressive episode, severe depressive episode, recurrent mild depressive episode, recurrent moderate depressive episode, recurrent severe depressive episode, recurrent depression without current symptoms and dysthymia, generalized anxiety disorder, antisocial personality disorder, anorexia nervosa, bulimia, binge eating disorder and ADHD.
* Having a family history of mental illness is assessed prior to treatment, screening for having a family history of dependence / substance abuse, bipolar disorder, depression, minor depression, neuropsychiatric condition, anxiety, panic disorder, psychosis, social anxiety disorder, social anxiety disorder-like symptoms, suicide attempts or suicide completed.
* Treatment process factors including perceived treatment credibility measured during the second week in treatment, measured with the Credibility/Expectancy Questionnaire (CEQ) where patients' attitudes to the credibility of the treatment and expectancy regarding treatment effectiveness are rated. Second, treatment adherence is measured at post-treatment, reflecting the degree of use of the ICBT program operationalized as the total number of activated treatment modules.

Measurements only administered at screening/pre-treatment:

* Patient Health Questionnare 9 (PHQ-9; all participants)
* Insomnia Severity Index (ISI; all participants)
* Liebowitz Social Anxiety Scale - (LSAS-SR; all participants)
* Panic Disorder Severity Scale - (PDSS-SR; all participants)
* Social Phobia Inventory (SPIN; all patients)
* The Alcohol Use Disorders Identification Test (AUDIT; all participants)
* The Drug Use Disorders Identification Test (DUDIT; all participants)
* The Adult Self Report Scale (ASRS-V1; all patients)

Behavioural measurements before/while undergoing MRI (all participants):

* Positive and Negative Affect Schedule (PANAS)
* Affect (valence and arousal). "How much pleasure or discomfort are you feeling right now? (1-9)" and "How calm or upset do you feel right now? (1-9)"
* Karolinska Sleepiness Scale (KSS)
* Subjective unit of discomfort (SUD): fear and distress (0-100)
* Self-rated health (SRH-7)
* Social Network Index (SNI)
* Short Grit Scale (SGI)

Predictors of treatment outcome

1. Behavioral predictor(s) of treatment outcome:

   * Questions about desired and expected treatment improvement. These include a) treatment credibility and b) modified PHQ-9, LSAS-SR and ISI questionnaires where the participants' expectation after completed treatment is self-rated for each item as well as participants' desire of improvement on a 0-100 scale for each item.
   * Ecological momentary assessments (EMA) with repeated sampling of participants' current behaviors and experiences in real time (4 times/day, during approximately 5 days prior to MRI procedure), including sleep problems, sleepiness, social anxiety, depressive symptoms, fear and discomfort. The purpose is to measure different and varied experiences / feelings over time. Variability in experiences will be compared to the participant's variability in brain function to answer the question of whether emotion variability can predict treatment outcomes. The specific EMA questions include the following: PHQ-2, Karolinska Sleepiness Scale (KSS), item 1 from ISI, item 11 and 15 from LSAS-SR and the subjective units of discomfort (fear and distress).
   * Emotion categorical ambiguity task
2. Brain-signal variability predictor(s), as derived from the following BOLD-fMRI experiments (all participants):

   * Face localizer task
   * Repetition suppression: faces (neutral, sad, angry, fear), scenes, verbal condition (á 60-90 seconds)
   * Faces
   * Scenes
   * Mooney faces
   * Retinotopy, i.e., traveling-wave method

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-5 criteria for depression, social anxiety or insomnia. Diagnosis and measures of symptom burden and functional level are made through a structured interview, the Mini-International Neuropsychiatric Interview (M.I.N.I.) and self-assessments of symptoms. Healthy controls should not be relevant to psychiatric treatment nor meet criteria for any psychiatric condition according to the M.I.N.I.
* Being able to read, write and speak Swedish in order to be able to read the treatment texts and be able to make phone calls.
* Having basic computer skills to be able to complete surveys via the Internet and access the treatment platform.

Exclusion Criteria:

* Physical or mental illnesses who are either contraindicated for treatment (for example, bipolar disorder that can be exacerbated by treatment) or for other reasons need other treatments (e.g. severe depression, suicidal behavior, psychotic illnesses or extensive cognitive difficulties).
* High alcohol consumption or other ongoing drug use.
* Answering "yes" to any of the following questions will be excluded for participation: 1) "Have you or have you had any electrical / battery operated implants in your body? For example, a pacemaker, medication pump, neurostimulator, hearing implant, or other electrical / battery controlled implant?" 2) "Have you done any surgery on the abdomen, chest, heart or brain, eyes, ears? For example, vessel clips, or objects such as screws, heart valve, shunt or prosthesis?" 3) "Do you have or have you had any metallic object in your body?" 4) "If a woman, are you pregnant or breastfeeding?" 5) "Do you undergo dialysis or have kidney dysfunction?" Participants who answer yes to these follow-up questions will be interviewed more closely to determine if MRI security can be guaranteed and whether the MRI signal will have significant disruptions, for example due to dental scaffolding. 1) "If you have any abdominal, thoracic, heart or brain, eyes, ears? Do you have any inoperable object that has ferromagnetic properties?" The patient will be asked to consult his doctor about this. 2) "If you have a dental rack, what type of dental rack (fixed or removable, metal plates / rails or wire)"?

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Reported in previous studies from the clinic:
  * Depression: mean age 37.9 (SD=11.8) yrs, 33% males, time since symptom debut, years 10.4 (SD=9.9), baseline MADRS-S scores 25.13 (SD=6.67); 72% on current psychotropic medication.
  * Insomnia: mean age 46.1 (SD=13.6) yrs, 70% males, baseline ISI scores 20.4 (SD=3.7); baseline MADRS-S score 25.5 (SD=6.8), 72% on current sleep medication 64%, on antidepressant medication 36%.
  * Social anxiety: mean age 32.51 (SD=8.98), 54% males, baseline LSAS-SR score 71.23 (SD=24.57), time since symptom debut, years 15.95 (SD=10.99), on current psychotropic medication 68% (SD=0.47).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Patient Health Questionnaire 9 - Self Assessment (PHQ-9) to Post-treatment | Up to 6 months
  The questionnaire has nine items. Overall score ranges from 0 to 27. Lower scores indicates a better outcome.
Change from Baseline Insomnia Severity Index - Self Assessment (ISI) to Post-treatment | Up to 6 months
  The questionnaire has seven items. The overall score ranges from 0 to 28. Lower scores indicates a better outcome.
Change from Baseline Liebowitz Social Anxiety Scale - Self Assessment (LSAS-SR) to Post-treatment | Up to 6 months
  The questionnaire has 48 items. The overall score ranges from 0 to 144. Lower scores indicates a better outcome.

SECONDARY OUTCOMES:
Consultation Satisfaction Questionnaire (CSQ-8) to Post-treatment | 3 months
  The questionnaire has 8 items. The overall score ranges from 8 to 32. Higher scores indicate a better outcome.
Social Phobia Inventory - Self Assessment (SPIN) 17 items. Overall score 0-68. | Up to 6 months
  Self Assessment, 17 items. Overall score 0-68. Lower scores indicates a better outcome.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Up to 6 months
  Self Assessment, 12 items. Overall score 0-100%. Lower scores indicate a better outcome.
Change from Baseline Generalized Anxiety Disorder Scale (GAD-7) to Post-treatment | Up to 6 months
  The questionnaire has seven items. The overall score ranges from 0 to 21. Lower scores indicate a better outcome.
Montgomery Åsberg Depression Rating Scale - Self Assessment (MADRS-S) | Up to 6 months
  Self Assessment, 9 items. Overall score 0-54. Lower scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer Kristoffer, PhD, Principal Investigator — Department of Clinical Neuroscience, Karolinska Institutet
Locations (1):
- Internetpsykiatri, Huddinge, Stockholm County, Sweden

REFERENCES:
- [Background] Schwiedrzik CM, Melloni L, Schurger A. Mooney face stimuli for visual perception research. PLoS One. 2018 Jul 6;13(7):e0200106. doi: 10.1371/journal.pone.0200106. eCollection 2018. PMID 29979727
- [Background] Wandell BA, Dumoulin SO, Brewer AA. Visual field maps in human cortex. Neuron. 2007 Oct 25;56(2):366-83. doi: 10.1016/j.neuron.2007.10.012. PMID 17964252
- [Background] Hariri AR, Mattay VS, Tessitore A, Kolachana B, Fera F, Goldman D, Egan MF, Weinberger DR. Serotonin transporter genetic variation and the response of the human amygdala. Science. 2002 Jul 19;297(5580):400-3. doi: 10.1126/science.1071829. PMID 12130784
- [Background] Wang S, Yu R, Tyszka JM, Zhen S, Kovach C, Sun S, Huang Y, Hurlemann R, Ross IB, Chung JM, Mamelak AN, Adolphs R, Rutishauser U. The human amygdala parametrically encodes the intensity of specific facial emotions and their categorical ambiguity. Nat Commun. 2017 Apr 21;8:14821. doi: 10.1038/ncomms14821. PMID 28429707
- [Background] Garrett DD, Kovacevic N, McIntosh AR, Grady CL. Blood oxygen level-dependent signal variability is more than just noise. J Neurosci. 2010 Apr 7;30(14):4914-21. doi: 10.1523/JNEUROSCI.5166-09.2010. PMID 20371811
- [Background] Garrett DD, Nagel IE, Preuschhof C, Burzynska AZ, Marchner J, Wiegert S, Jungehulsing GJ, Nyberg L, Villringer A, Li SC, Heekeren HR, Backman L, Lindenberger U. Amphetamine modulates brain signal variability and working memory in younger and older adults. Proc Natl Acad Sci U S A. 2015 Jun 16;112(24):7593-8. doi: 10.1073/pnas.1504090112. Epub 2015 Jun 1. PMID 26034283
- [Background] Mansson KN, Frick A, Boraxbekk CJ, Marquand AF, Williams SC, Carlbring P, Andersson G, Furmark T. Predicting long-term outcome of Internet-delivered cognitive behavior therapy for social anxiety disorder using fMRI and support vector machine learning. Transl Psychiatry. 2015 Mar 17;5(3):e530. doi: 10.1038/tp.2015.22. PMID 25781229
- [Background] Hedman E, Ljotsson B, Kaldo V, Hesser H, El Alaoui S, Kraepelien M, Andersson E, Ruck C, Svanborg C, Andersson G, Lindefors N. Effectiveness of Internet-based cognitive behaviour therapy for depression in routine psychiatric care. J Affect Disord. 2014 Feb;155:49-58. doi: 10.1016/j.jad.2013.10.023. Epub 2013 Oct 26. PMID 24238951
- [Background] Blom K, Jernelov S, Kraepelien M, Bergdahl MO, Jungmarker K, Ankartjarn L, Lindefors N, Kaldo V. Internet treatment addressing either insomnia or depression, for patients with both diagnoses: a randomized trial. Sleep. 2015 Feb 1;38(2):267-77. doi: 10.5665/sleep.4412. PMID 25337948
- [Background] Hedman E, Andersson E, Ljotsson B, Axelsson E, Lekander M. Cost effectiveness of internet-based cognitive behaviour therapy and behavioural stress management for severe health anxiety. BMJ Open. 2016 Apr 25;6(4):e009327. doi: 10.1136/bmjopen-2015-009327. PMID 27113231
- [Background] Mansson KNT, Waschke L, Manzouri A, Furmark T, Fischer H, Garrett DD. Moment-to-Moment Brain Signal Variability Reliably Predicts Psychiatric Treatment Outcome. Biol Psychiatry. 2022 Apr 1;91(7):658-666. doi: 10.1016/j.biopsych.2021.09.026. Epub 2021 Oct 12. PMID 34961621